CLINICAL TRIAL: NCT03381456
Title: Task-dependent Operation of a Mechanism Intracortical Inhibition in Dystonia
Acronym: LICIdystonie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013_51; 2014-A00244-43 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Dystonia, Primary
MeSH Terms: conditions — Dystonic Disorders

STUDY DESIGN:
Intervention Model Description: 10 patient with dystonia and 10 healthy subject paired by sex and age.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy subject (Experimental): LICI
  Interventions: Other: LICI
- Dystonic subject (Experimental): LICI
  Interventions: Other: LICI

INTERVENTIONS:
Other: LICI — Paired pulse TMS to measure LICI and late cortical disinhibition

SUMMARY:
Cortical excitability depends on inhibitory mechanisms efficiency among which long latency intracortical inhibition (LICI) can be studied by paired pulses transcranial magnetic stimulation (TMS). Some recent evidences suggest that LICI may be one of the mechanisms by which the motor comment is adapted to the ongoing motor task with LICI strength being dependent on task complexity. In writer cramp and musician cramp, two forms of dystonia, the cortical excitability is not correctly modulated in some complex gestures. the hypothesis is that this task dependent perturbation of excitability in writer cramp could be due to a lack of LICI efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patient with hand dystonia : writers cramp
* Subject affiliated to social security regimen.

For healthy volunteers :

* Healthy volunteer without neurological disorders based on sensorimotor examination.
* Subject affiliated to social security regimen.

Exclusion Criteria :

* Subject unable to receive informed consent (dementia).
* Contraindication to Transcranial Magnetic Stimulation(TMS) (epilepsia, intracranial metalic foreign object, hearing device, cochlear implant).
* Patient using a psychotrope treatment.
* Patient under guardianship or curatorship.
* Pregnant or nursing women.
* Patient with a cardiac stimulator.

For healthy volunteers only :

• Abnormal neurological evaluation based on sensorimotor examination or neurological history ( epilepsy, stroke ; brain or spinal cord surgery ; history of neurological disease affective sensitive and motor control)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
long-interval intracortical inhibition (LICI) level | Baseline
  Amount of inhibition at interstimulus intervals of between 50 to 300ms

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Derambure, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No